CLINICAL TRIAL: NCT03856580
Title: Developing Tailored Delivery and Adherence Interventions for Use of Long-acting Biomedical HIV Prevention Strategies by Transgender Women
Brief Title: Long-acting Biomedical HIV Prevention in Transgender Women
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: New York State Psychiatric Institution-wide research pause affecting all studies
Sponsor: University of Colorado, Denver (Other)
Collaborators: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-3620tx
Record Dates: First submitted 2019-02-22; First posted 2019-02-27 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: HIV Prevention; Transgender Women

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Self-injection (Experimental): Participants will be trained on how to self-inject (intramuscular, gluteal muscle) an inert version of injectable cabotegravir. The inert substance is intended to mimic injectable cabotegravir as closely as possible (e.g., injection equipment, location of injection, volume of injection is identical to injectable cabotegravir). Specifically, participants will self-inject their choice of 300mg vitamin B12 or saline (3ml fluid) every 2 months for a total of 6 months (for a total of 4 injections). Participants will complete interviews and brief surveys on their experience. Additionally, they will be given access to an mHealth app to improve adherence, which will contain informational content such as instructions on how to self-inject, FAQs about self-injection, study contact information, etc..
  Interventions: Behavioral: Alternative long-acting PrEP injection strategies; Behavioral: mHealth adherence app
- Injection by HCP at "drop-in" clinics (Experimental): Participants will report to a "drop-in" clinic, where a healthcare provider will inject them with an inert version of injectable cabotegravir. "Visits will take <10 minutes, and participants will be able to come whenever they want (when their injection is due) during clinic "drop-in" hours, which will be staggered in 2-hour windows during each week day. The inert substance that will be injected is intended to mimic injectable cabotegravir as closely as possible (described above). Participants will complete interviews and brief surveys on their experience. Additionally, they will be given access to an mHealth app to improve adherence, which will contain informational content such as "drop-in" clinic hours, directions to the "drop-in" clinic site, study contact information, etc...
  Interventions: Behavioral: Alternative long-acting PrEP injection strategies; Behavioral: mHealth adherence app
- Control group (No Intervention): Participants will make an appointment when their injection is due to report to our clinic to complete injections. Visits and the injection protocol will follow similar procedures to HPTN-083/084. Participants will not have access to the mHealth adherence app.

INTERVENTIONS:
Behavioral: Alternative long-acting PrEP injection strategies — Participants in the two intervention groups will complete injection procedures (e.g., self-injection, injection by healthcare providers at "drop-in" clinics) to determine if this could facilitate improved adherence to an inert version of long-acting cabotegravir injections
  Arms: Injection by HCP at "drop-in" clinics; Self-injection
Behavioral: mHealth adherence app — Participants in the two experimental arms will be given a smartphone application, designed to facilitate adherence (this app will be developed during earlier phases of the study using in-depth interviews and "design session" groups)
  Arms: Injection by HCP at "drop-in" clinics; Self-injection

SUMMARY:
Transgender women (TW) have unique challenges related to HIV prevention medication adherence. Left unaddressed, these challenges will prevent TW from accessing the promising long-acting HIV prevention tools in the development pipeline. This study will develop a replicable process to tailor the delivery of these tools and an adherence intervention (that will include an mHealth app) to the needs of TW, using the example of inert injectable cabotegravir. Work builds on a pilot study to identify tailored methods to deliver injectable cabotegravir in TW, such as self-injection and injection by a healthcare provider at at "drop-in" clinic. The investigators will use qualitative methods (e.g., interviews, group discussions called "Design Sessions") to design the adherence intervention and the mHealth app. Then, investigators will execute a partially randomized patient-preference trial to determine if TW are able to use tailored injection strategies (self-injection or injection by a healthcare provider at "drop-in clinics") to improve adherence, compared to a control group of TW who will engage a protocol based on HPTN-083/084. This will serve as a "proof of concept" for the future R01 that will test this on a larger scale. Research and training will take place at NYSPI/Columbia, in affiliation with, 1) Project AFFIRM, a study of transgender identity (R01HD079603; PI: Bockting), that will provide infrastructure for critical research activities (e.g., recruitment), and 2) SLAP-HIV, a clinical trial to produce a long-acting form of cabotegravir (e.g., injection; UM1 AI120184; PI: Hope). SLAP-HIV will provide clinical oversight (e.g., ensure tailored delivery strategies are feasible).

ELIGIBILITY:
Inclusion Criteria:

* HIV-negative
* self-identified transgender woman (or woman assigned male at birth)
* at least 18 years old
* willing to complete injections
* own a smartphone that uses apps
* speak English or Spanish
* willing to take an HIV test
* live in the NYC/tri-state area
* report receptive or penetrative genital-to-genital sex with another person in the last 3 months

Exclusion Criteria:

* HIV-positive
* does not identify as a transgender woman (or woman assigned male at birth)
* younger than 18
* unwilling to complete injections
* does not own a smartphone that uses apps
* does not speak English or Spanish
* refuses HIV test
* lives outside of the NYC/tri-state area
* has not had receptive or penetrative genital-to-genital sex with another person in the last 3 months

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Assigned male at birth but identifies as a woman, Transgender woman, Woman of transgender experience
Enrollment: 19 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Number of completed injections at month 6 | 6 months
  Number of completed injections by each of the possible intervention arms (self-injection, injection by HCP at "drop-in" clinics), compared to the controls group at month 6.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Rael, Ph.D., Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute/Columbia University Medical Center, New York, New York, United States